CLINICAL TRIAL: NCT05441163
Title: ProActIF-01 Trial: Feasibility Study of an Individualized Program of Nutrition and Adapted Physical Activity in Frail Patients With Advanced Digestive Cancers
Acronym: ProActIF-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IC 2021-01
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: CANCER
Keywords: gastrointestinal cancer
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms | interventions — Glutamyl Aminopeptidase; Diet Therapy

STUDY DESIGN:
Intervention Model Description: Intervention : standard of care plus a supervised 8-week combined APA and nutrition individualized program
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APA and nutrition program (Experimental)
  Interventions: Other: APA and nutrition intervention

INTERVENTIONS:
Other: APA and nutrition intervention — - APA intervention: weekly supervised sessions at home with the APA professional combined with unsupervised sessions, alone or with the APA partner, for 8 weeks.
  The supervised session will be broken down as follows: warm-up block (approximately 10'), aerobic block (15'), muscle strengthening/resistance block (15') and stretching/relaxation block (10'). The remaining 10' will be used to review the session and the individual sessions. This program can be adapted to the needs and abilities of the patient if necessary.
  - Nutritional intervention: dietitian weekly visits at home during 8 weeks with dietetic counseling; decision of oral, enteral and/or parenteral feeding validated by the clinical steering committee according to the Société Francophone de Nutrition Clinique et Métabolisme (SFNCM) guidelines.

SUMMARY:
The ProActIF-01 trial aims to assess the feasibility of a supervised 8-week combined APA and nutrition individualized program, in advanced digestive cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Age ≥ 18 years (no superior limit), men and women.
3. First-line treatment (chemotherapy and/or immunotherapy) for advanced disease (previous adjuvant therapy allowed).
4. Histologically confirmed adenocarcinoma or squamous cell carcinoma of digestive tract (colorectal, esogastric, pancreas, biliary tract).
5. Locally advanced or metastatic disease not amenable to surgery, radiation, or combined modality therapy with curative intent (previous resection of primary tumor allowed).
6. ECOG PS 0-2. Note: patient with ECOG PS 3-4 are excluded because they are usually not eligible for chemotherapy.
7. Having at least one risk factor among the following: ECOG PS = 2 and/or malnutrition (weight loss ≥5% of body weight in 1 month or ≥10% in 6 months or compared to usual weight before disease or BMI <18.5 kg/m2 for patients aged <70 years and 22 for patients aged ≥70 years).
8. Life expectancy ≥ 8 weeks.
9. Able to answer questionnaires in French.
10. Availability of an APA partner (family member or friend who will attend the exercise sessions at least once a week).
11. Registration in a national health care system (Couverture Maladie Universelle, CMU included).

Exclusion Criteria:

1. Neuroendocrine carcinoma histology.
2. Any medical (including psychiatric, musculoskeletal, or neurological) condition contra-indicating exercise practice.

   Note: bone or brain metastases are allowed if not at risk of complications and if associated symptoms do not limit exercise practice; radiotherapy is allowed if terminated ≥ 2 weeks prior to study inclusion.
3. Nonfunctional gastrointestinal tract compromising oral/enteral feeding. Note: gastrointestinal tract obstruction is allowed if the tumor can be bypassed or stented (e.g. esophageal cancer with gastric tube-stoma or esophageal stent).
4. Participation to another physical activity or nutritional structured intervention program (in the first two months).

   Note: participation to another concomitant clinical trial (except for trials evaluating supportive care programs involving physical activity or nutritional intervention) is allowed but the patient must inform the Investigator and get an authorization from the Sponsor.
5. Major risk of refeeding syndrome: BMI <16 kg/m2 or low blood levels of potassium, phosphorus or magnesium prior to refeeding (Note : oral and/or IV supplementation is allowed and patients can be included after correction of blood levels of potassium, phosphorus and magnesium).

   Note : - malnourished patients who have started nutritional intervention (ONS, artificial nutrition) are eligible if they have not started chemotherapy/immunotherapy.

   - progressive increase in calory/protein is possible in severely malnourished patients but the targets should be reached before the 2nd chemotherapy/immunotherapy cycle.
6. Pregnancy or breastfeeding.
7. Protected adults (individuals under guardianship by court order).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2027-02-08 (Estimated); Study Completion 2028-04-08 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of a supervised 8-week combined APA and nutrition individualized program | 8 weeks
  The rate of eligible and evaluable patients who complete successfully the nutrition and APA program. For a given patient, the success of the program is defined by:
  * at least 75% of the planned supervised APA sessions: 6 of 8 home-based sessions with an APA professional
  * at least 75% of the nutritional evaluations: 6 of 8 planned home-based evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, MD, Principal Investigator — Institut Curie Saint-Cloud
Locations (17):
- France (17):
  - CHRU de Tours, Tours, Institut Curie
  - Institut du cancer Avignon-Provence, Avignon
  - Institut Bergonié, Bordeaux
  - Centre de Lutte Contre le Cancer Jean Perrin, Clermont-Ferrand
  - Institut Daniel Hollard - Groupe Hospitalier Mutualiste, Grenoble
  - centre Oscar Lambret, Lille
  - Hôpital de la Croix Rousse - Hospices Civils de Lyon, Lyon
  - centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier (ICM), Montpellier
  - Institut Curie, Paris
  - Hôpital COCHIN AP-HP, Paris
  - CHU Reims, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - Institut de Cancérologie de l'Ouest (ICO), Saint-Herblain
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).